CLINICAL TRIAL: NCT01733238
Title: PNT2258-02: A Pilot Phase II Study of PNT2258 for Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Study of PNT2258 for Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNT2258-02
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: PNT2258; Lymphoma; Non-Hodgkin's Lymphoma; NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — PNT100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PNT2258 (Experimental): PNT2258 120 mg/m2 will be administered as a 2-hour intravenous infusion on days 1-5 of a 21-day cycle. Treatment may continue (unless there is disease progression or the occurrence of unacceptable toxicity) for a total of 6 cycles of therapy.
  Interventions: Drug: PNT2258

INTERVENTIONS:
Drug: PNT2258

SUMMARY:
This study is sponsored by Sierra Oncology, Inc. formerly ProNAi Therapeutics, Inc. It study is a multi-center, nonrandomized, open-label, pilot Phase II investigation of PNT2258 to characterize anti-tumor activity and collect safety data on patients with relapsed or refractory lymphoma.

DETAILED DESCRIPTION:
PNT2258 will be administered at a dose of 120 mg/m2, as a 3-hour intravenous (IV) infusion on days 1-5 of a 21-day cycle. Treatment may continue (unless there is disease progression or the occurrence of unacceptable toxicity) for a total of 6 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the patient.
2. Participants must be ≥18 years of age.
3. Morphologically confirmed diagnosis of non-Hodgkin's lymphoma (NHL).
4. At least a single measureable tumor mass (long axis > 1.5 cm).
5. An FDG-PET positive baseline scan.

   a. A positive scan is defined per revised Cheson criteria as "focal or diffuse FDG uptake above background in a location incompatible with normal anatomy or physiology, without a specific standardized uptake value cutoff".
6. Disease that has relapsed after administration of primary therapy that included:

   1. Rituximab and
   2. CHOP, EPOCH, bendamustine or similar chemotherapy or subsequent salvage regimen.

   Note: Relapse is defined as progression after a complete response to therapy or radiographic evidence of active disease after a partial response or stable disease.
7. Have received three or fewer complete courses of systemic cytotoxic regimens. Note: Rituximab (alone or in combination with cytotoxic chemotherapy) is not considered a cytotoxic regimen.
8. No previous exposure to PNT2258.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
10. Have discontinued all prior anti-cancer therapies for at least 21 days; biologic therapy for at least 4 half-lives of the drug(s); radio-immunotherapy (10 weeks); autologous stem cell transplantation (SCT) (3 months) and must be at a stable baseline regarding any acute toxicity associated with prior therapy.
11. Adequate organ function including:

    1. Hematologic Function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L prior to treatment. Platelets ≥ 100 x 109/L.
    2. Hepatic: Total Bilirubin ≤ 1.5 x ULN and serum transaminase levels ≤ 2.5 x upper limits of normal (ULN).
    3. Renal: Serum creatinine ≤2 x ULN or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with serum creatinine levels above 2x ULN.

Exclusion Criteria:

1. Candidates for HDT and autologous SCT. Note: Patients who progressed > 3 months after high-dose therapy (HDT)/SCT are eligible.
2. Concurrent malignancies requiring treatment.
3. Symptomatic central nervous system (CNS) or leptomeningeal involvement of lymphoma.
4. Concurrent serious medical conditions (as determined by the Principal Investigator) including, but not limited to, HIV-associated lymphoma; active bacterial, fungal or viral infections.
5. Signs and symptoms of heart failure characterized as greater than New York Heart Association (NYHA) Class I.
6. History of myocardial infarct or prolonged corrected QT (QTc) interval (>450 milliseconds (msecs) for males or >470 msecs for females) or other significant cardiac abnormalities.
7. Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Klencke, M.D., Study Chair — Sierra Oncology LLC - a GSK company; Ayad Al-Katib, MD, Principal Investigator — St. John Hospital and Medical Center, Van Elslander Cancer Center
Locations (3):
- United States (3):
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Cancer and Hematology Centers of Western Michigan, P.C., Grand Rapids, Michigan
  - St. John Hospital and Medical Center, Van Elslander Cancer Center, Grosse Pointe Woods, Michigan

REFERENCES:
- [Derived] Harb W, Lakhani NJ, Messmann R, Klencke B, Al-Katib AM. A Phase 2 Study of PNT2258 for Treatment of Relapsed or Refractory B-Cell Malignancies. Clin Lymphoma Myeloma Leuk. 2021 Dec;21(12):823-830. doi: 10.1016/j.clml.2021.07.016. Epub 2021 Jul 23. PMID 34417162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in November 2012 and the first subject was enrolled on 22 January 2013. A total of 15 subjects were screened. Subjects were enrolled at oncology clinics in the USA.
Groups:
- PNT2258: PNT2258 120 mg/m2 administered on days 1-5 of a 21-day cycle.
Period: Overall Study
Arm/Group | PNT2258
Started | 13
Completed (8 subjects completed the Induction Phase and 7 subjects started Maintenance Phase) | 8 (8 subjects completed the Induction Phase and 7 subjects started Maintenance Phase)
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: All patients who passed the screening in the study
Arm/Group | PNT2258
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: Years] | 65.0 [40.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Subjects who had a best response of complete response or partial response as assessed by the investigator
Time Frame: 39 months
Population: All subjects who received at least 1 dose of PNT2258
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PNT2258
Number analyzed (Participants) | 13
percentage of participants | 53.8 [25.1 to 80.8]

2. Secondary Outcome: Progression-free Survival
Description: The time from Cycle 1 Day 1 until the date of lymphoma progression or death from any cause, or to the last date at which progression status was adequately assessed for censored observation
Time Frame: 39 months
Population: All subjects who received at least 1 dose of PNT2258
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PNT2258
Number analyzed (Participants) | 13
months | 9.5 [2.4 to 32.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until 30 days after the last dose of PNT2258 for each subject
Arm/Group | PNT2258
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrilation (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anticoagulation drug level above therapeutic (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=13)
Nausea (Gastrointestinal disorders) | 12
Chills (General disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 8
Headache (Nervous system disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 6
Dizziness (Nervous system disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Hypertension (Vascular disorders) | 6
Insomina (Psychiatric disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Pain (General disorders) | 6
Pyrexia (General disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Fall (Injury, poisoning and procedural complications) | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Asthenia (General disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Oedema peripheral (General disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eyelid oedema (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diverticulum (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival cyst (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Lip disorder (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Salivary gland mass (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Application site erythema (General disorders) | 1
Chest pain (General disorders) | 1
Device occlusion (General disorders) | 2
Gait disturbance (General disorders) | 1
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 2
Infusion site erythema (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Infusion site oedema (General disorders) | 1
Infusion site pain (General disorders) | 1
Local swelling (General disorders) | 1
Localised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Performance status decreased (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 2
Tongue injury (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Blood phosphorus increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Breath sounds abnormal (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Electrocardiogram repolarisation abnormality (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypermetabolism (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Areflexia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes